CLINICAL TRIAL: NCT05502016
Title: Family Model Diabetes Self-Management Education in Faith-Based Organizations in the Republic of the Marshall Islands
Brief Title: Family Model DSME in FBOs in the RMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 263202; 1R01DK128145-01A1 (NIH)
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Palliative Care; Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Family model diabetes self-management education and support
  Interventions: Behavioral: Family Model Diabetes Self-Management Education and Support
- Wait-list Control (Active Comparator): Family model diabetes self-management education and support
  Interventions: Behavioral: Family Model Diabetes Self-Management Education and Support (Wait-list)

INTERVENTIONS:
Behavioral: Family Model Diabetes Self-Management Education and Support — Participants assigned to this arm receive an intervention that includes a culturally adapted family model diabetes self-management education and support with at least one participating family member in a faith-based organization setting.
  Arms: Intervention
Behavioral: Family Model Diabetes Self-Management Education and Support (Wait-list) — Participants assigned to this arm will wait approximately 12 weeks to receive an intervention that includes a culturally adapted family model diabetes self-management education and support with at least one participating family member in a faith-based organization setting.
  Arms: Wait-list Control

SUMMARY:
Health disparities in the Republic of the Marshall Islands are striking, with extremely high rates of type 2 diabetes. Documented prevalence of type 2 diabetes in the Marshall Islands ranges from 20%-50%.This is significantly higher than the global (8.5%) and United States (11%) prevalence. Diabetes doubles the risk of heart disease; is the leading cause of kidney failure, lower limb amputation, and acquired blindness; and reduces life expectancy by as much as 15 years. Diabetes self-management education and support is critical for persons with diabetes. This study aims to conduct a cluster-randomized controlled trial using a wait-list control to evaluate the effectiveness of family model diabetes self-management education and support when delivered in faith-based organizations (i.e., churches) in Marshallese by trained community health workers. The study will be conducted with up to 288 participants with type 2 diabetes and up to 288 of their family members. The primary study outcome will be glycemic control as measured by HbA1c. Secondary biometric measures include: fasting glucose, weight, body mass index, and blood pressure. Survey data will be collected pre-intervention, immediately post-intervention, four months post-intervention, and 12 months post-intervention for the intervention arm of the study. The control arm of the study will have two pre-intervention data collections before beginning the intervention. Data will then be collected from the control group immediately post-intervention, four months post-intervention, and 12 months post intervention.

ELIGIBILITY:
Inclusion Criteria:

* self-reported Marshallese
* 18 years of age or older
* have type 2 diabetes (defined as having HbA1c equal to or greater than 6.5%)
* have at least one family member willing to take part in the study

Exclusion Criteria:

* has received diabetes self-management education in the past five years
* has a condition that makes it unlikely that the participant will be able to follow the protocol, such as terminal illness, non-ambulatory, severe mental illness, severely impaired vision or hearing, eating disorder
* plans to move out of the geographic region

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic control, measured by change in mean HbA1c (%) from baseline | Baseline, Immediate post-intervention, 4 months post-intervention, 12 months post-intervention
  Point of care tests will be utilized to calculate HbA1c levels for each participant. The primary outcome measure is change in mean HbA1c (%) from baseline to immediate post-intervention, 4 months post-intervention, and 12 months post-intervention. Analyses will be adjusted for baseline HbA1c, sex, age, education, marital status, employment status, use of diabetes medications, and clustering of participants within churches.

CONTACTS AND LOCATIONS:
Overall Officials: Pearl McElfish, PhD, Principal Investigator — University of Arkansas
Locations (1):
- UAMS Institute for Community Health Innovation, Springdale, Arkansas, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT05502016/ICF_000.pdf